CLINICAL TRIAL: NCT01450241
Title: Short-term Antibiotic Treatment for Unexplained Fever in Solid Cancer Patients With Febrile Neutropenia: Randomized-controlled Trial
Brief Title: Short-term Antibiotic Treatment for Unexplained Fever in Solid Cancer Patients With Febrile Neutropenia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment, no funding
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, leibovici leonard, Professor, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RabinMC6249
Record Dates: First submitted 2011-09-17; First posted 2011-10-12 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Febrile Neutropenia
Keywords: Febrile neutropenia; Unexplained fever; Duration; Short-term antibiotic treatment
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early antibiotic discontinuation (Experimental): Antibiotic treatment stopped after 72h, regardless of fever.The antibiotics used will be piperacillin tazobactam for high-risk patients and amoxycillin-clavulanate + ciprlofloxacin for low-risk patients (defined by MASCC scoring system). Alternatives in case of penicillin allergy will be ceftazidine and levofloxacin, respectively.
  Interventions: Other: Early antibiotic discontinuation
- Usual practice (Other): Antibiotic treatment continued according to accepted guidelines and current clinical practice. The antibiotics used will be piperacillin tazobactam for high-risk patients and amoxycillin-clavulanate + ciprlofloxacin for low-risk patients (defined by MASCC scoring system). Alternatives in case of penicillin allergy will be ceftazidine and levofloxacin, respectively.
  Interventions: Other: Usual practice

INTERVENTIONS:
Other: Early antibiotic discontinuation — Antibiotic treatment for unexplained febrile neutropenia stopped after 72 hours, regardless of fever
  Arms: Early antibiotic discontinuation
Other: Usual practice — Continued antibiotic treatment as accepted by guidelines for febrile neutropenia
  Arms: Usual practice

SUMMARY:
The purpose of this study is to determine whether short-course antibiotic therapy is safe and effective for the treatment of cancer patients with febrile neutropenia.

DETAILED DESCRIPTION:
Febrile neutropenia remains a major cause of morbidity in solid cancer patients. There is an unresolved question regarding the appropriate duration of antibiotic treatment for patients with febrile neutropenia of unknown origin. Current guidelines recommend at least seven days of antibiotic treatment. Several studies have demonstrated the safety of early antibiotic discontinuation in patients with febrile neutropenia. We plan an open label randomized controlled trial to compare early antibiotic discontinuation to the accepted prolonged antibiotic treatment protocol

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years providing signed informed consent
* Patients with solid tumors, lymphoma, multiple myeloma or chronic lymphocytic leukemia, regardless of disease status or previous chemotherapy
* Documented febrile neutropenia
* No clinically or microbiologically documented infection after 72 hours

Exclusion Criteria:

* Previous enrollment in this study
* Concurrent participation in another interventional trial
* Severe sepsis or septic shock
* Acute leukemia, autologous or allogeneic hematopoietic stem-cell transplantation
* Diarrhea suspected by treating physician to be Irinotecan induced
* Any antibiotic treatment for >48h in the last week before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of all-cause mortality, severe infection, severe diarrhea or fever | After day 7 from randomization until day 30
  Composite outcome of all-cause mortality, severe infection (defined as clinically or microbiologically documented infection with systemic inflammatory response syndrome (SIRS)), severe diarrhea (>=3 daily for >=2 days) or fever (>38)
Total febrile or antibiotic days | From the day of randomization until day 30
  Total febrile or antibiotic days from the day of randomization until day 30, defined as a day with one or more temperature measurement >38.0°C or a day on which antibiotic treatment was prescribed for any reason other than prophylaxis

SECONDARY OUTCOMES:
Clinically and/or microbiologically documented infections | 30 days
  Clinically and/or microbiologically documented infections within 30 days of randomization. We will use the 2008 CDC/NHSN surveillance definitions of health-care associated infections for bacterial infections (including Clostridium difficile) and the 2008 revised definitions for invasive fungal infections.
Total in-hospital days | 30 days
  Total in-hospital days from the day of randomization up to day 30
Re-admission | 30 days
  Rates of re-admission for any reason other than planned chemotherapy.
Antibiotic treatment | After day 7 from randomization until day 30
  Patients receiving antibiotic treatment after day 7 from randomization until day 30
Antifungal treatment | 30 days
  Institution of antifungal treatment
Duration of intravenous antibiotic treatment | 30 days
  Duration of intravenous antibiotic treatment
Duration of neutropenia | 30 days
  Duration of neutropenia
Development of resistance | 30 days
  Development of resistance, defined as clinical isolates resistant to antibiotics previously used in the febrile episode. Surveillance sampling will not be conducted.
All-cause mortality | 30 days
  All-cause mortality
Infection-related mortality | 30 days after randomization
  Cause of death adjudicated by the trial's safety committee

CONTACTS AND LOCATIONS:
Overall Officials: Mical Paul, MD, Principal Investigator — Rabin Medical Center; Leonard Leibovici, Prof, Principal Investigator — Rabin Medical Center; Dafna Yahav, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Beilinson Hospital, Petah Tikvah, Israel